CLINICAL TRIAL: NCT01595451
Title: Brain Mechanisms of Acupuncture Treatment in Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Massachusetts General Hospital (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Robert Edwards, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2011P000757
Record Dates: First submitted 2012-05-08; First posted 2012-05-10 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Chronic Low Back Pain; Low Back Pain; Back Pain
Keywords: Acupuncture; Back Pain; Lower Back Pain; Brigham and Women's Hospital; Massachusetts General Hospital; Effects of Acupuncture
MeSH Terms: conditions — Low Back Pain; Back Pain | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Traditional Acupuncture (Active Comparator): Acupuncture will be delivered to 12 points traditionally used to treat chronic low back pain.
  Interventions: Procedure: Acupuncture
- Non-traditional Acupuncture (Placebo Comparator): You will receive non-traditional acupuncture at 12 points for chronic low back pain.
  Interventions: Procedure: Acupuncture

INTERVENTIONS:
Procedure: Acupuncture — A licensed acupuncturist will perform acupuncture for six, 30 minute treatment sessions.

SUMMARY:
We are doing this study to investigate the effects of acupuncture on chronic low back pain. We are interested in learning about brain activity during pain. We plan to look at brain activity at the beginning and the end of the study, after 6 sessions of acupuncture treatment. You will be randomly assigned to one of two groups to receive either real or placebo acupuncture.

Acupuncture has been used for many years to help relieve pain. However, it is not clear how acupuncture works. Acupuncture may relieve pain by changing activity in the nervous system. Some studies indicate that acupuncture may relieve the low back pain. However, we need more research to see how well acupuncture works to relieve pain for people with this condition.

In this study, we will measure your brain activity before and after you do exercises to make your back pain worse. We will also measure your brain activity while inflating a pressure cuff device on your lower leg. We will measure this brain activity using a research tool called functional MRI (fMRI). Functional MRI is a very fast MRI that uses radio waves and a magnet, and allows the study investigators to look at changes in blood flow to different parts of the brain when there are changes in brain activity.

ELIGIBILITY:
Inclusion Criteria:

* Meet the Classification Criteria of the chronic LBP (having low back pain for more than 6 months), as determined by the referring physician.
* Subjects must be able to provoke or exacerbate their cLBP using our calibrated exercise-like maneuver.
* At least 4/10 clinical pain on the 11-point LBP severity scale on average during the past two weeks prior to enrollment.
* At least a 10th grade English-reading level; English can be a second language provided that the patients feel they understand all the questions used in the assessment measures.
* Right handed individuals
* Must have had a prior evaluation of their low back pain by a health care provider, which may include radiographic studies. Documentation of this evaluation will be obtained from subject's medical record.

Exclusion Criteria:

* Specific causes of back pain (e.g., cancer, fractures, spinal stenosis, infections)
* Complicated back problems (e.g., prior back surgery, medico-legal issues)
* Possible contraindications for acupuncture (e.g., coagulation disorders, cardiac pacemakers, pregnancy, seizure disorder), and conditions that might confound treatment effects or interpretation of results (e.g., severe fibromyalgia, rheumatoid arthritis)
* Conditions making treatment difficult (e.g., paralysis, psychoses, or other severe psychiatric problems based on the judgment of a physician investigator and/or a T score >60 on the psychological assessments performed during Session 1)
* Prior acupuncture treatment for back pain; 1 year minimum for any other condition.
* The intent to undergo surgery during the time of involvement in the study.
* History of cardiac, respiratory, or nervous system disease that, in the judgment of a physician investigator, precludes participation in the study because of a heightened potential for adverse outcome (e.g., asthma, claustrophobia)
* Presence of any contraindications to MRI scanning (e.g., cardiac pacemaker, metal implants, fear of closed spaces, pregnancy)
* Active substance abuse disorders within the last 24 months, based on subject self-report
* Unresolved medical legal/disability/workers compensation claims
* Radicular knee pain extending below the knee
* Use of more than 60 mg morphine equivalent prescription opioids or steroids for pain.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 79 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Pain improvement in patients with lower back pain | 6 week study
  Acupuncture in patients with lower back pain

CONTACTS AND LOCATIONS:
Overall Officials: Robert Edwards, Ph.D., Principal Investigator — Brigham and Women's Hospital
Locations (1):
- MGH - Martinos Center, Charlestown, Massachusetts, United States